CLINICAL TRIAL: NCT00891982
Title: A Phase 3B, Multicenter, Assessor-Blinded Study of the Tolerability of Clindamycin 1%-Tretinoin 0.025% Gel Used in Conjunction With Benzoyl Peroxide 4% Wash in Subjects With Mild to Moderate Facial Acne Vulgaris
Brief Title: A Clinical Study to Evaluate the Tolerability of a Topical Antibiotic and Retinoid Used in a Combined Regimen With a BPO Wash
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114679
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin, tretinoin drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTGel plus BPO wash (Experimental): Benzoyl peroxide (BPO) Wash in the morning and CTGel in the evening
  Interventions: Drug: CTGel/ BPO Wash
- CTGel (Active Comparator): Soap Free Cleanser in the morning and CTGel in the evening
  Interventions: Drug: Soap Free Cleanser and CTGel

INTERVENTIONS:
Drug: CTGel/ BPO Wash — Benzoyl Peroxide (BPO) wash will be used once daily in the morning for 28 days
  Clindamycin and Tretinoin (CT) gel will be used once daily in the evening for 28 days.
  Other Names: Veltin
  Arms: CTGel plus BPO wash
Drug: Soap Free Cleanser and CTGel — Soap Free Cleanser will be used once daily in the morning for 28 days
  Clindamycin and Tretinoin gel will be used once daily in the evening for 28 days.
  Other Names: Veltin
  Arms: CTGel

SUMMARY:
The purpose of this study is to evaluate the tolerability of a combined regimen of a topical antibiotic and retinoid and a benzoyl peroxide wash.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild to moderate facial acne vulgaris, with no history of known or suspected hypersensitivity or previous allergic reaction to any of the ingredients of the study products (eg, topical antibiotics, retinoids or benzoyl peroxide), capable of understanding and willing to provide signed and dated written voluntary informed consent and able to complete the study and to comply with study instructions.
* Female subjects of childbearing potential must have a negative urine pregnancy test result at baseline and practice a reliable method of contraception throughout the study.

Exclusion Criteria:

* Use of topical antibiotics on the face within the past 2 weeks or use of systemic antibiotics within the past 4 weeks.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - Dermatology Associates Research, Coral Gables, Florida
  - Grekin Skin Institute, Warren, Michigan
  - Dermatology Consulting Services, High Point, North Carolina
  - The Skin Wellness Center, PC, Knoxville, Tennessee
  - Premier Clinical Research, Spokane, Washington

REFERENCES:
- [Background] Draelos ZD, Potts A, Alio Saenz AB; W0265-306 Study Group. Randomized tolerability analysis of clindamycin phosphate 1.2%-tretinoin 0.025% gel used with benzoyl peroxide wash 4% for acne vulgaris. Cutis. 2010 Dec;86(6):310-8. PMID 21284283

RESULTS

PARTICIPANT FLOW:
Groups:
- CTGel Plus BPO Wash: BPO Wash in the morning and CTGel in the evening
Period: Overall Study
Arm/Group | CTGel Plus BPO Wash | CTGel
Started | 30 | 31
Completed | 28 | 30
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTGel Plus BPO Wash | CTGel | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Customized [Number; unit: participants]
  <18 years | 16 | 14 | 30
  Between 18 and 45 years | 14 | 17 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 24 | 26 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 2 | 3 | 5
  White | 24 | 28 | 52
  More than one race | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61
ISGA [Number; unit: participants] — Investigator's Static Global Assessment measured on a 6 point scale where 0=normal, clear skin; 1 = skin almost clear; 2 = Some noninflammatory lesions are present, with few inflammatory lesions; 3 = Noninflammatory lesions predominate, with multiple inflammatory lesions evident; 4 = Inflammatory lesions are more apparent: many comedones and papules/pustules,there may or may not be a few nodulocystic lesions; and 5=highly inflammatory lesions predominate.
  participants
    Grade 2 | 9 | 11 | 20
    Grade 3 | 18 | 15 | 33
    Grade 4 | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Local Tolerability - Skin Dryness
Description: Local tolerability and irritation potential based on investigator assessments of dryness, scaling, and erythema in the areas of study product application. Grading will use the following scale:
  0 - None
  1. - Trace
  2. - Mild
  3. - Moderate
  4. - Marked
  5. - Severe
Time Frame: Screening/baseline
Measure: Number; unit: participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
participants
  Grade 0 | 28 | 26
  Grade 1 | 2 | 4
  Grade 2 | 0 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 0 | 0

2. Primary Outcome: Local Tolerability - Skin Dryness
Description: as for outcome 1
Time Frame: Week 1
Measure: Number; unit: participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
participants
  Grade 0 | 12 | 16
  Grade 1 | 5 | 8
  Grade 2 | 5 | 5
  Grade 3 | 6 | 0
  Grade 4 | 0 | 1
  Grade 5 | 1 | 0
  Missing | 1 | 1

3. Primary Outcome: Local Tolerability - Skin Dryness
Description: as for outcome 1
Time Frame: Week 2
Measure: Number; unit: participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
participants
  Grade 0 | 15 | 17
  Grade 1 | 7 | 8
  Grade 2 | 5 | 4
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 2

4. Primary Outcome: Local Tolerability - Skin Dryness
Description: as for outcome 1
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
participants
  Grade 0 | 19 | 19
  Grade 1 | 7 | 11
  Grade 2 | 2 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 0

5. Primary Outcome: Local Tolerability - Skin Scaling
Description: as for outcome 1
Time Frame: Screening/baseline
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 29 | 28
  Grade 1 | 1 | 2
  Grade 2 | 0 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 0 | 0

6. Primary Outcome: Local Tolerability - Skin Scaling
Description: as for outcome 1
Time Frame: Week 1
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 13 | 19
  Grade 1 | 5 | 5
  Grade 2 | 5 | 3
  Grade 3 | 5 | 2
  Grade 4 | 1 | 1
  Grade 5 | 0 | 0
  Missing | 1 | 1

7. Primary Outcome: Local Tolerability - Skin Scaling
Description: as for outcome 1
Time Frame: Week 2
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 17 | 19
  Grade 1 | 6 | 6
  Grade 2 | 4 | 4
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 2

8. Primary Outcome: Local Tolerability - Skin Scaling
Description: as for outcome 1
Time Frame: Week 4
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 20 | 25
  Grade 1 | 6 | 5
  Grade 2 | 2 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 0

9. Primary Outcome: Local Tolerability - Erythema (Redness)
Description: as for outcome 1
Time Frame: Screening/baseline
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 22 | 22
  Grade 1 | 4 | 4
  Grade 2 | 1 | 4
  Grade 3 | 3 | 1
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 0 | 0

10. Primary Outcome: Local Tolerability - Erythema (Redness)
Description: as for outcome 1
Time Frame: Week 1
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 10 | 18
  Grade 1 | 8 | 5
  Grade 2 | 8 | 2
  Grade 3 | 3 | 3
  Grade 4 | 0 | 2
  Grade 5 | 0 | 0
  Missing | 1 | 1

11. Primary Outcome: Local Tolerability - Erythema (Redness)
Description: as for outcome 1
Time Frame: Week 2
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 17 | 12
  Grade 1 | 5 | 9
  Grade 2 | 5 | 6
  Grade 3 | 1 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 2

12. Primary Outcome: Local Tolerability - Erythema (Redness)
Description: as for outcome 1
Time Frame: Week 4
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 15 | 16
  Grade 1 | 5 | 9
  Grade 2 | 4 | 4
  Grade 3 | 4 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 0

13. Secondary Outcome: Subject Assessment of Burning/Stinging
Description: Each symptom will be graded by the subject based upon the subject's impression during the previous week using the following scale:
  0 - None
  1. - Trace
  2. - Mild
  3. - Moderate
  4. - Marked
  5. - Severe
Time Frame: Screening/baseline
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 27 | 26
  Grade 1 | 2 | 1
  Grade 2 | 1 | 3
  Grade 3 | 0 | 0
  Grade 4 | 0 | 1
  Grade 5 | 0 | 0
  Missing | 0 | 0

14. Secondary Outcome: Subject Assessment of Burning/Stinging
Description: as for outcome 13
Time Frame: Week 1
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 14 | 15
  Grade 1 | 7 | 8
  Grade 2 | 3 | 3
  Grade 3 | 5 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 1
  Missing | 1 | 2

15. Secondary Outcome: Subject Assessment of Burning/Stinging
Description: as for outcome 13
Time Frame: Week 2
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 22 | 15
  Grade 1 | 5 | 12
  Grade 2 | 1 | 2
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 2

16. Secondary Outcome: Subject Assessment of Burning/Stinging
Description: as for outcome 13
Time Frame: Week 4
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 23 | 14
  Grade 1 | 4 | 15
  Grade 2 | 0 | 1
  Grade 3 | 0 | 1
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 3 | 0

17. Secondary Outcome: Subject Assessment of Itching
Description: as for outcome 13
Time Frame: Screening/Baseline
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 25 | 21
  Grade 1 | 3 | 6
  Grade 2 | 2 | 2
  Grade 3 | 0 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 0 | 0

18. Secondary Outcome: Subject Assessment of Itching
Description: as for outcome 13
Time Frame: Week 1
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 13 | 14
  Grade 1 | 6 | 9
  Grade 2 | 8 | 6
  Grade 3 | 2 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 1 | 2

19. Secondary Outcome: Subject Assessment of Itching
Description: as for outcome 13
Time Frame: Week 2
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 18 | 18
  Grade 1 | 6 | 10
  Grade 2 | 3 | 1
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 2 | 2

20. Secondary Outcome: Subject Assessment of Itching
Description: as for outcome 13
Time Frame: Week 4
Measure: Number; unit: Participants
Arm/Group | CTGel Plus BPO Wash | CTGel
Number analyzed (Participants) | 30 | 31
Participants
  Grade 0 | 18 | 21
  Grade 1 | 9 | 8
  Grade 2 | 0 | 2
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Missing | 3 | 0

ADVERSE EVENTS:
Arm/Group | CTGel Plus BPO Wash | CTGel
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 1/30 | 5/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTGel Plus BPO Wash (N=30) | CTGel (N=31)
Application site dryness (General disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.